CLINICAL TRIAL: NCT05888194
Title: The Effect of Mucogyne® Gel on Wound Healing
Acronym: ARTHEMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUCG-233
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Perineal Tear and Episiotomy

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mucogyne group (Experimental): In Mucogyne group, each eligible patient will receive a box of Mucogyne® gel. The patient will apply Mucogyne® gel, 48-hours after delivery, everyday, twice a day, massaging it into the intimate area, for a 10-day period.
  Interventions: Device: Mucogyne® gel
- Control group (No Intervention): Standard of care e.i no treatment

INTERVENTIONS:
Device: Mucogyne® gel — In Mucogyne group, each eligible patient will receive a box of Mucogyne® gel. The patient will apply Mucogyne® gel, 48-hours after delivery, everyday, twice a day, massaging it into the intimate area, for a 10-day period.
  Arms: Mucogyne group

SUMMARY:
The aim of this post-market clinical follow up study is to confirm the efficacy and safety of topical application of Mucogyne® gel in the process of wound healing, when used in accordance with its approved labeling, in the context of postpartum perineal wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women with singleton pregnancy
2. Have a perineal tear or mediolateral episiotomy
3. First (with cutaneous injury) and 2nd-degree perineal tear/episiotomy, whose length and depth are as the following:

   * depth (from the fourchette into the greatest depth of the perineal body) ≤3cm,
   * length of vaginal mucosa (from the fourchette to the apex of the vaginal tear) ≤4cm
   * length of skin (from the fourchette along perineal skin towards the anus) ≤3cm
4. Is able to understand the study related information and to give a written informed consent,
5. Has signed the informed consent form before beginning any study procedure,
6. Has no condition that may interfere with the study assessments,
7. Is able to comply with protocol requirements and respect the conditions of the study,
8. Accept to come to the mentioned hospital 12(+/-2) days after childbirth
9. Affiliated to the Social Security system

Exclusion Criteria:

1. Postpartum complications, or developed early bleeding after delivery
2. Third and fourth degree perineal tear.
3. Previous vaginal/perineal surgery within the year preceding the inclusion in the study
4. Had undergone extended episiotomy (incision size > 3 - 4 cm)
5. Anal fissures.
6. Known hypersensitivity to any of the medical device ingredients
7. With local infectious lesions in the area to be repaired.
8. Who use drugs known to disturb wound healing (example : anticoagulants during pregnancy (based on self-reports))
9. Had a history of diseases known to disturb wound healing (e.g. systemic, heart, and renal diseases, coagulation disorders, immune deficiency, connective tissue disorders, diabetes, anemia (with hemoglobin level < 9 g/dl) and hemophilia)
10. Immunosuppressive treatment.
11. Heavy cigarettes smoker (i.e., more than 15 cigarettes or equivalent/day, according to the mothers and their documented records),
12. Patients under legal protection or under guardianship and patients deprived of freedom
13. Has any other severe chronic or acute medical or psychiatric condition that in the judgment of the Investigator, could interfere with the study assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of topical application of Mucogyne® gel in postpartum perineal wound healing promotion. | Day 0 to Day 12 (+/-2) after delivery
  Wound healing will be assessed using the perineal healing scale after episiotomy or perineal tear, the Redness, Oedema, Ecchymosis, Discharge, Approximation (REEDA) scale, change between baseline (48h postpartum) and 12 days postpartum days (after 10 days of application of Mucogyne® gel) will be calculated.The REEDA scale is an observational check list used for assessing perineal wound healing that was primarily developed by Davidson (1974). It can be used to assess all types of postpartum perineal trauma. It has five components namely Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges. Each component takes a score ranged from 0 to 3. Total REEDA score ranges between 0 and 15. Higher score indicates poor wound healing while lower score indicates good wound healing. The total score of REEDA scale was categorized as follows; Completely healed from 0 to 2, Moderately healed from 3 to 5, Mildly healed from 6 to 8, and Not healed from 9 to 15.

SECONDARY OUTCOMES:
To describe wound characteristics | Day 0 to Day 12 (+/-2) after delivery
  Wound characteristics will be described using the Redness, Oedema, Ecchymosis, Discharge, Approximation (REEDA) scale sub-score at each visit. The REEDA scale is an observational check list used for assessing perineal wound healing that was primarily developed by Davidson (1974). It can be used to assess all types of postpartum perineal trauma. It has five components namely Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges. Each component takes a score ranged from 0 to 3. Total REEDA score ranges between 0 and 15. Higher score indicates poor wound healing while lower score indicates good wound healing. The total score of REEDA scale was categorized as follows; Completely healed from 0 to 2, Moderately healed from 3 to 5, Mildly healed from 6 to 8, and Not healed from 9 to 15.
To assess pain relief (related to the vaginal wound) | Day 0 to Day 12 (+/-2) after delivery
  The presence of perineal pain (related to the vaginal wound) at rest, in movement, while sitting, while urinating and defecating
To assess the need/use of pain relieving drugs | Day 0 to Day 12 (+/-2) after delivery
  Number of used pain-relieving drug related to the vaginal wound healing
To assess change in clinical status | Day 0 to Day 12 (+/-2) after delivery
  Change in clinical status will be assessed by Clinical Global Impressions scale, (CGI-I). The CGI was developed for use in clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.
To assess change in clinical status | Day 0 to Day 12 (+/-2) after delivery
  Change in clinical status will be assessed by Patients' Global Impression of Change scale (PGIC). The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
To assess the patient wound cosmetic appearance | Day 0 to Day 12 (+/-2) after delivery
  Wound cosmetic appearance will be assessed using a scale from the "worst scar" to the "best scar"
To assess the overall patient's satisfaction | Day 0 to Day 12 (+/-2) after delivery
  Patient satisfaction will be assessed using Patient Satisfaction Score (PSS) rated based on scores of 0 to 10, with higher scores indicating better satisfaction and lower scores indicating poorer satisfaction.
To assess re-appropriation and acceptance of the body by the patient | Day 0 to Day 12 (+/-2) after delivery
  Re-appropriation and acceptance of the body will be assessed by a questionnaire. The body reappropriation scale is composed of 5 questions in 7 points with 1="Strongly agree" and 7="Strongly disagree". This scale looks at the patient's ability to look at her scar in a mirror, to clean it, to touch it and to massage it. One question concerns the impact of the scar's appearance on the patient's self-esteem.
To assess the patient perception of the Medical Device | Day 0 to Day 12 (+/-2) after delivery
  A customized questionnaire about sensory analysis of the study product (texture, ease of spreading, softness after application, aqueous, freshness, etc.)
To assess compliance with the Medical Device use | Day 0 to Day 12 (+/-2) after delivery
  Number of days of use
To assess the safety of Mucogyne® gel : Number, nature and characteristics of any incident reported: incidence, seriousness, severity, resolution. | Day 0 to Day 12 (+/-2) after delivery

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Lille, Lille
  - CHU Montpellier, Montpellier
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No